CLINICAL TRIAL: NCT06756516
Title: Effect of Feldenkrais Method on Balance in Patients With Mechanical Low Back Pain: A Randomized Controlled Trial
Brief Title: Effect of Feldenkrais Method on Balance in Patients With Mechanical Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Mohamed Emad Fahmy Mohamed, Teaching assistant Biomechanics department, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005554
Record Dates: First submitted 2024-12-23; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Mechanical Low Back Pain
Keywords: Feldenkrais method; mechanical low back pain; balance
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feldenkrais Method balance exercises (Experimental): Balance exercises in Feldenkrais method plus core stability exercises
  Interventions: Other: Feldenkrais Method and Core stabilization
- Core stability exercises only (Active Comparator): Core strengthening exercises to engage global and local stabilizers of the spinal column as Bridging exercises, Side bridging exercise, plank, side plank, McGill Abdominal exercises.
  Each exercise will be repeated for 3 sets with 8 repetitions with hold for 5 seconds.
  Interventions: Other: Core stability exercises

INTERVENTIONS:
Other: Feldenkrais Method and Core stabilization — Balance exercises from supine lying position using Feldenkrais style, plus core stabilization exercises.
  Arms: Feldenkrais Method balance exercises
Other: Core stability exercises — trunk deep muscles activation and engaging using exercises as bridging, side bridging, plank, side plank and McGill Abdominal
  Arms: Core stability exercises only

SUMMARY:
The goal of this clinical trial is to learn if Feldenkrais method affects balance in patients with mechanical low back pain. The main questions it aims to answer is:

does Feldenkrais method affects balance in patients with mechanical low back pain.

Participants will:

Be assessed for inclusion using slump and straight leg raise tests. Visit the clinic twice every week for sessions. Assessed pre and post treatment using Biodex Balance.

DETAILED DESCRIPTION:
Sample size calculation showed that our sample is 40. Forty patients with mechanical low back pain not referring beyond the knee will be recruited from Souad Kafafi Hospital and multiple outpatient clinics in Giza, Egypt. Inclusion criteria is male or female patients, 18-45 years, mechanical pain for the last 6 months, with no previous surgeries or diseases in the spine. Treatment strategy include 10 treatment sessions for each allocated subject. Core strengthening exercises and Feldenkrais method (balance exercises) are the treatment approached used in this study. Two experienced physical therapists will apply the treatment in the Faculty of Physical therapy clinic. Overall, mediolateral, and anteroposterior stability will be assessed for each patient. The measurement will be done twice pretreatment and immediately after the last session.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical back pain.
* Symptoms lasted for the last 6 months.
* Not referring beyond the knee.
* Mild to moderate pain in Numerical Pain Rating Scale and mild to moderate disability on Oswestry Disability Index

Exclusion Criteria:

* Spine Surgeries
* Chronic diseases
* Accidents and Fractures

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-05-14 (Estimated); Study Completion 2025-05-28 (Estimated)

PRIMARY OUTCOMES:
Balance | Baseline and 5 weeks.
  Using Biodex Balance System 3 parameters will be assessed. Overall stability Mediolateral stability Anteroposterior stability

CONTACTS AND LOCATIONS:
Overall Officials: Neveen A Abdelraouf, Professor, Study Chair — Cairo University Faculty of Physical Therapy; Aya A Khalil, Lecturer, Study Director — Cairo University Faculty of Physical Therapy; Shereen M Said, Lecturer, Study Director — Misr University for Science and Technology; Mohamed E Fahmy, Instructor, Principal Investigator — Misr University for Science and Technology
Locations (1):
- Misr University for Science and Technology, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be shared by the principal investigator using email address mohamed.khater@must.edu.eg upon request.
Supporting Information: Study Protocol
Time Frame: After the date of publication of this work by 3 months.
Access Criteria: The requests will be assessed by the principal investigator. The data will be sent by the formal email address.